CLINICAL TRIAL: NCT04689191
Title: A Randomized, Double-Blind, Controlled, Non-inferiority Phase III Trial of a Group A and C Meningococcal Polysaccharide Vaccine in Healthy Children Aged 2-6 Years
Brief Title: A Phase III Clinical Trial of the Group A and C Meningococcal Polysaccharide Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Cun (Unknown)
Collaborators: Yunnan Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor-Investigator, Wei Cun, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20190702
Record Dates: First submitted 2020-12-08; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Meningitis, Meningococcal
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Vaccine (Experimental): One dose of Experimental Group A and C meningococcal polysaccharide vaccine
  Interventions: Biological: Experimental Group A and C meningococcal polysaccharide vaccine
- Active Comparator Vaccine (Active Comparator): One dose of Control Group A and C meningococcal polysaccharide vaccine
  Interventions: Biological: Control Group A and C meningococcal polysaccharide vaccine

INTERVENTIONS:
Biological: Experimental Group A and C meningococcal polysaccharide vaccine — One dose of Experimental Group A and C meningococcal polysaccharide vaccine
  Arms: Experimental Vaccine
Biological: Control Group A and C meningococcal polysaccharide vaccine — One dose of Control Group A and C meningococcal polysaccharide vaccine
  Arms: Active Comparator Vaccine

SUMMARY:
This study is a randomized, double-blinded, and controlled phase III clinical trial of the Group A and C meningococcal polysaccharide vaccine to evaluate the safety and immunogenicity of the vaccine in healthy infants aged 2-6 years.

DETAILED DESCRIPTION:
This study was divided into two stages. The first stage study was an early safety assessment study among 80 subjects. The first stage study was conducted gradually in 20 subjects aged 18-50 years, 20 subjects aged 7-17 years, and 40 subjects aged 2-6 years. The second phase was a randomized, double-blind, controlled, non-inferiority phase III clinical trial in 1200 healthy infants aged 2-6 years, to evaluate the immunogenicity and safety of the experimantal vaccine after immunization.

ELIGIBILITY:
* The First stage study (An early safety assessment study):
* 18-50 years group:

  * Inclusion Criteria:

    1. Healthy adults aged 18 to 50 years.
    2. Proven legal identity.
    3. Participants should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
    4. Participants should be able to communicate well with investigators, understand and comply with the requirements of this trial.
    5. Axillary temperature ≤37.0℃.
  * Exclusion Criteria:

    1. Contraindications for vaccination.
    2. History of allergy to vaccines or drugs.
    3. History of Epidemic Cerebrospinal Meningitis.
    4. Immunization with any Group A meningococcal conjugate vaccine or polysaccharide vaccine within 12 months.
    5. Immunization with any Group A and C meningococcal conjugate vaccine or polysaccharide vaccine within 3 years.
    6. Immunization with any vaccine within 30 days.
    7. Patients with convulsion, epilepsy, encephalopathy and psychiatric history or family history of epilepsy.
    8. History of abnormal clinical manifestations and serious diseases to be excluded, including but not limited to nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, bones and other system diseases, and a history of malignant tumors.
    9. Those who developed acute disease or acute attack of chronic disease.
    10. Surgical removal of spleen or other important organs for any reason.
    11. History of thrombocytopenia or other coagulation disorders may cause contraindication of subcutaneous injection.
    12. Blood products such as immunoglobulin were received within 30 days before vaccination.
    13. Have received immunosuppressive therapy or other immunomodulatory drugs within 6 months before signing the informed consent form (Note: inhaled or topical hormone drugs, except those with an interval of 14 days or more from the date of signing the informed consent form).
    14. Those who participated in other clinical studies.
    15. Participants who have a positive pregnancy test, or are breastfeeding, or plan to become pregnant, or plan to donate sperm or eggs from the screening to 12 months after the second vaccination.
    16. Any other situations judged by investigators as not suitable for participating in this study.
* 7-17 years group:

  * Inclusion Criteria

    1. Healthy volunteer aged 7 to 17 years.
    2. Proven legal identity.
    3. Participants and their legal guardians should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
    4. Participants and their legal guardians should be able to communicate well with investigators, understand and comply with the requirements of this trial.
    5. Axillary temperature ≤37.0℃.
  * Exclusion Criteria:

    1. Contraindications for vaccination.
    2. History of allergy to vaccines or drugs.
    3. History of Epidemic Cerebrospinal Meningitis.
    4. Immunization with any Group A meningococcal conjugate vaccine or polysaccharide vaccine within 12 months.
    5. Immunization with any Group A meningococcal conjugate vaccine or polysaccharide vaccine within 3 years.
    6. Immunization with any vaccine within 30 days.
    7. Patients with convulsion, epilepsy, encephalopathy and psychiatric history or family history of epilepsy.
    8. Participant who has congenital heart disease, congenital malformation, Down's syndrome, sickle cell anemia or severe diseases with previous clinical manifestations that need to be excluded, including but not limited to nervous system, genetic defect disease (such as faba bean disease), cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bone system diseases, and History of malignant tumor.
    9. Those who developed acute disease or acute attack of chronic disease.
    10. Surgical removal of spleen or other important organs for any reason.
    11. History of thrombocytopenia or other coagulation disorders may cause contraindication of subcutaneous injection.
    12. Blood products such as immunoglobulin were received within 30 days before vaccination.
    13. Have received immunosuppressive therapy or other immunomodulatory drugs within 6 months before signing the informed consent form (Note: inhaled or topical hormone drugs, except those with an interval of 14 days or more from the date of signing the informed consent form).
    14. Those who participated in other clinical studies.
    15. Women with positive pregnancy test after menarche.
    16. Any other situations judged by investigators as not suitable for participating in this study.
* 2-6 years group:

  * Inclusion Criteria

    1. Healthy children aged 2 to 6 years.
    2. Proven legal identity.
    3. Participants' legal guardians should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
    4. Participants' legal guardians should be able to communicate well with investigators, understand and comply with the requirements of this trial.
    5. Axillary temperature ≤37.0℃.
  * Exclusion Criteria:

    1. Contraindications for vaccination.
    2. History of allergy to vaccines or drugs.
    3. History of Epidemic Cerebrospinal Meningitis.
    4. Immunization with any Group A and C meningococcal conjugate vaccine or polysaccharide vaccine.
    5. Immunization with any Group A meningococcal conjugate vaccine or polysaccharide vaccine within 12 months.
    6. They were vaccinated with live attenuated vaccine within 14 days before vaccination and subunit or inactivated vaccine within 7 days (copy of vaccination certificate of subjects);
    7. Participants with convulsion, epilepsy, encephalopathy and psychiatric history or family history of epilepsy.
    8. Participant who has congenital heart disease, congenital malformation, Down's syndrome, sickle cell anemia or severe diseases with previous clinical manifestations that need to be excluded, including but not limited to nervous system, genetic defect disease (such as faba bean disease), cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bone system diseases, and History of malignant tumor.
    9. Those who developed acute disease or acute attack of chronic disease.
    10. Surgical removal of spleen or other important organs for any reason.
    11. History of thrombocytopenia or other coagulation disorders may cause contraindication of subcutaneous injection.
    12. Blood products such as immunoglobulin were received within 30 days before vaccination.
    13. Have received immunosuppressive therapy or other immunomodulatory drugs within 6 months before signing the informed consent form (Note: inhaled or topical hormone drugs, except those with an interval of 14 days or more from the date of signing the informed consent form).
    14. Those who participated in other clinical studies.
    15. Any other situations judged by investigators as not suitable for participating in this study.

The Second stage study (A phase III clinical trial )

* Inclusion Criteria

  1. Healthy children aged 2 to 6 years.
  2. Proven legal identity.
  3. Participants' legal guardians should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
  4. Participants' legal guardians should be able to communicate well with investigators, understand and comply with the requirements of this trial.
  5. Axillary temperature ≤37.0℃.
* Exclusion Criteria:

  1. Contraindications for vaccination.
  2. History of allergy to vaccines or drugs.
  3. History of Epidemic Cerebrospinal Meningitis.
  4. Immunization with any Group A and C meningococcal conjugate vaccine or polysaccharide vaccine.
  5. Immunization with any Group A meningococcal conjugate vaccine or polysaccharide vaccine within 12 months.
  6. They were vaccinated with live attenuated vaccine within 14 days before vaccination and subunit or inactivated vaccine within 7 days (copy of vaccination certificate of subjects);
  7. Participants with convulsion, epilepsy, encephalopathy and psychiatric history or family history of epilepsy.
  8. Participant who has congenital heart disease, congenital malformation, Down's syndrome, sickle cell anemia or severe diseases with previous clinical manifestations that need to be excluded, including but not limited to nervous system, genetic defect disease (such as faba bean disease), cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bone system diseases, and History of malignant tumor.
  9. Those who developed acute disease or acute attack of chronic disease.
  10. Surgical removal of spleen or other important organs for any reason.
  11. History of thrombocytopenia or other coagulation disorders may cause contraindication of subcutaneous injection.
  12. Blood products such as immunoglobulin were received within 30 days before vaccination.
  13. Have received immunosuppressive therapy or other immunomodulatory drugs within 6 months before signing the informed consent form (Note: inhaled or topical hormone drugs, except those with an interval of 14 days or more from the date of signing the informed consent form).
  14. Those who participated in other clinical studies.
  15. Any other situations judged by investigators as not suitable for participating in this study.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1280 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate of Group A meningococcal bactericidal antibody | 28 days after vaccination
  Seroconversion rate of Group A meningococcal bactericidal antibody at day 28 after vaccination
Seroconversion rate of Group C meningococcal bactericidal antibody | 28 days after vaccination
  Seroconversion rate of Group C meningococcal bactericidal antibody at day 28 after vaccination

SECONDARY OUTCOMES:
Adverse reactions/events rate | 7 days after vaccination
  Occurence of adverse reactions/events after vaccination
Adverse reactions/events rate | 28 days after vaccination
  Occurence of adverse reactions/events after vaccination
Serious adverse events | 6 months after the second vaccination
  Occurence of Serious adverse events after vaccination
GMT of Group A meningococcal bactericidal antibody | 28 days after the second vaccination
  GMT of Group A meningococcal bactericidal antibody at day 28 after the second vaccination
GMT of Group C meningococcal bactericidal antibody | 28 days after the second vaccination
  GMT of Group C meningococcal bactericidal antibody at day 28 after the second vaccination

OTHER OUTCOMES:
GMT of IgG antibody against Hepatitis A | 28 days after the second vaccination
  GMT of IgG antibody against Hepatitis A at day 28 after vaccination
Seropositive rate of IgG antibody against Hepatitis A | 28 days after the second vaccination
  Seropositive rate of IgG antibody against Hepatitis A at day 28 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, Mater, Principal Investigator — Yunnan Center for Disease Control and Prevention
Locations (1):
- Yunnan Center for Disease Control and Prevention, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No